CLINICAL TRIAL: NCT06895837
Title: Acute Effect of Exercise on Appetite, Appetite-Regulatory Hormones, and Energy Intake During Energy Restriction in Healthy Men
Brief Title: Effect of Exercise on Appetite in Response to Meals During Energy Restriction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Northern Border University (Other)
Responsible Party: Principal Investigator, James Dorling, PhD, Lecturer in Human Nutrition (Medicine), University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 200240250
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The participants will not perform any exercise and will receive 100% of their estimated energy needs.
- Severe-energy restriction (Experimental): The participants will not perform any exercise and will receive 25% of their estimated energy needs.
  Interventions: Other: Severe-energy restriction
- Severe-energy restriction with exercise (Experimental): The participants will run on the treadmill for 30 minutes and receive 25% of their estimated energy needs.
  Interventions: Other: Severe-energy restriction with exercise

INTERVENTIONS:
Other: Severe-energy restriction — The participants will receive only 25% of their estimated energy needs.
  Arms: Severe-energy restriction
Other: Severe-energy restriction with exercise — The participants will run on the treadmill for 30 minutes and receive 25% of their estimated energy needs.
  Arms: Severe-energy restriction with exercise

SUMMARY:
This study's primary aim is to investigate the acute effect of an exercise bout (30 minutes) on appetite and appetite-regulatory hormone responses during energy restriction. The researchers will also test if the exercise bout influences ad libitum energy intake after a period of energy restriction.

The researchers will compare three groups (control, severe-energy restriction, and severe-energy restriction with exercise) to see if exercise bout, during energy restriction, affects appetite, appetite-regulatory hormones, and energy intake in healthy men.

DETAILED DESCRIPTION:
Before the main experiments are conducted, participants will attend a screening visit where the participants will provide consent and complete questionnaires that assess their health, food preferences, and physical activity levels. Researchers will then measure the participants' height, weight, waist circumference, and body composition.

Once the eligibility criteria are confirmed, participants will participate in two treadmill tests to establish their maximum oxygen uptake (V̇O2 max).

After the screening visit, participants will participate in three main experiments, each lasting 24 hours: control, severe energy restriction, and severe energy restriction with exercise. These experiments will be conducted in a counterbalanced design. Each experiment will start around 9:30 AM, following an overnight fast of at least 10 hours. Participants will have a prescribed meal in the evening before each main experiment. After this meal, the participants are only allowed to drink water until the start of the main experiments.

During the exercise trial, participants will begin by running on a treadmill for 30 minutes at a speed estimated to achieve 75% of their V̇O2 peak, followed by a rest period in the laboratory. The same protocol will be followed in the control and severe-energy trials, except that no exercise will be performed. Participants will rest in the laboratory during both the control and energy-restricted trials. In the control trial, the participants will receive 100% of their estimated energy needs; in the energy-restricted trials, the participants will receive only 25%.

The participants will have standardized breakfast and lunch meals at 1h and 5h, respectively. At 24h, participants will be provided an ad libitum buffet meal in a private eating room.

The researchers will assess appetite ratings in each experiment using 100 mm visual analog scales. The researchers will also collect blood samples to analyze ghrelin, peptide YY (PYY), glucagon-like peptide 1 (GLP-1), and potentially other blood-borne measures.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 years or older.
* Have stable body mass for at least six months (within ±2 kg).

Exclusion Criteria:

* Females
* People who are younger than 18 or older than 65 years old.
* Following a special diet (e.g. weight loss, vegetarian or vegan, etc.).
* Have food allergies related to the study.
* Have significant contraindications to exercise (e.g., an injury that would inhibit running).
* Smoking.
* Taking any medications.
* Suffering from metabolic health issues, e.g., history of diabetes, cardiovascular disease, or eating disorders.
* Have any mental health conditions.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 14 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Peptide-YY (PYY) | At 0 (baseline), 0.5, 1, 1.5, 2, 3, 4, 5, 5.5, 6, 6.5, 7, and 23 hours
  The researchers will draw blood samples at different time points during the trial to measure the change in PYY blood levels. Area under the plasma concentration versus time curve (AUC) of PYY will be calculated using the trapezoidal rule.
Change in Ghrelin | At 0 (baseline), 0.5, 1, 1.5, 2, 3, 4, 5, 5.5, 6, 6.5, 7, and 23 hours
  The researchers will draw blood samples at different time points during the trial to measure the change in ghrelin blood levels. Area under the plasma concentration versus time curve (AUC) of ghrelin will be calculated using the trapezoidal rule.
Change in Glucagon-Like Peptide-1 (GLP-1) | At 0 (baseline), 0.5, 1, 1.5, 2, 3, 4, 5, 5.5, 6, 6.5, 7, and 23 hours
  The researchers will draw blood samples at different time points during the trial to measure the change in GLP-1 blood levels. Area under the plasma concentration versus time curve (AUC) of GLP-1 will be calculated using the trapezoidal rule.
Change in subjective appetite sensations | At 0 (baseline), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, 6, 6.5, 7, 23, 24, and 25 hours
  The researchers will assess the subjective appetite sensations using 100 mm visual analog scales (VAS) to measure appetite sensations (hunger, satiety, fullness, prospective food consumption, and desire to eat). The VAS are 100 mm long, with words anchored at each end expressing the most positive and negative ratings. Scores for each appetite construct range from 0-100.

SECONDARY OUTCOMES:
Energy Intake | At 24 hours
  To determine the amount of each food item consumed, the researchers will measure the difference in weight between before and after the meal. The researchers will use manufacturer details to determine energy consumption.
Macro-nutrient Intake | At 24 hours
  To determine the amount of each food item consumed, the researchers will measure the difference in weight between before and after the meal. The researchers will use manufacturer details to determine macro-nutrient consumption.

CONTACTS AND LOCATIONS:
Overall Officials: James Dorling, PhD, Principal Investigator — University of Glasgow
Locations (1):
- New Lister Building, Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The stored data will be pseudonymous and follow the guidelines of the General Data Protection Regulation enforced in May 2018. Hard copies of participant information forms, including consent forms and dietary intake records, will be kept in locked filing cabinets. Keys to the filing cabinets will only be available to the primary investigator. All databases will be password protected and stored on a university computer with firewalls.
  Participants' identifiable data will be stored in a locked cabinet. Digital data will be stored anonymously within the server of the University of Glasgow.
  This project's Principal Investigator will be responsible for sharing the research data.
  Data will be preserved in Enlighten, the official online repository of Glasgow University's research output.
Time Frame: Data will be preserved for 10 years.

REFERENCES:
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749
- [Background] Broom DR, Miyashita M, Wasse LK, Pulsford R, King JA, Thackray AE, Stensel DJ. Acute effect of exercise intensity and duration on acylated ghrelin and hunger in men. J Endocrinol. 2017 Mar;232(3):411-422. doi: 10.1530/JOE-16-0561. Epub 2016 Dec 20. PMID 27999089